CLINICAL TRIAL: NCT00685646
Title: A Phase III, Multicenter, Randomized, Controlled Study of Maximum Androgen Blockade With vs. Without Zoledronic Acid in Prostatic Cancer Patients With Metastatic Bone Disease
Brief Title: Androgen Blockade Therapy With or Without Zoledronic Acid in Treating Patients With Prostate Cancer and Bone Metastases
Acronym: ZAPCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIGU0705; KYUH-TRIGU0705 (Other: National Cancer Institute)
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: bone metastases; stage IV prostate cancer
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Androgen Antagonists; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive maximum androgen-blockade therapy and zoledronic acid for up to 24 courses.
  Interventions: Drug: antiandrogen therapy; Drug: zoledronic acid
- Arm II (Active Comparator): Patients receive maximum androgen-blockade therapy for up to 24 courses.
  Interventions: Drug: antiandrogen therapy

INTERVENTIONS:
Drug: antiandrogen therapy — Up to 24 courses of therapy
Drug: zoledronic acid — Up to 24 courses of therapy
  Arms: Arm I

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Androgen blockade therapy may lessen the amount of androgens made by the body. Zoledronic acid may help relieve some of the symptoms caused by bone metastasis. It is not yet known whether androgen-blockade therapy is more effective with or without zoledronic acid in treating patients with prostate cancer that has spread to the bone.

PURPOSE: This randomized phase III trial is studying androgen-blockade therapy given together with zoledronic acid to see how well it works compared with androgen-blockade therapy alone in treating patients with prostate cancer and bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the time to treatment failure in prostatic cancer patients with metastatic bone disease receiving maximum androgen-blockade therapy with vs without zoledronic acid.
* Evaluate the time to first skeletal-related events in these patients.
* Evaluate the overall survival of these patients.
* Evaluate the extent of disease on bone scan in these patients.
* Evaluate the pain scale and FACES pain-rating scale in these patients.
* Evaluate the safety of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive maximum androgen-blockade therapy and zoledronic acid for up to 24 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive maximum androgen-blockade therapy for up to 24 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with definitive diagnosis of prostatic cancer by histopathological diagnosis or cytology
* Androgen blockade therapy-, systemic chemotherapy-, bisphosphonates-naïve prostatic cancer patients
* Patients who are sensitive to androgen blockade therapy
* Patients with bone metastasis on bone scan (EOD ≥ 1)
* Patients who have Eastern Cooperative Oncology Group performance status (ECOG: 0-2)
* Patients who have prostate-specific antigen performance status (PSA ≧30 ng/mL)
* Patients who demonstrate appropriate bone marrow, hepatic and renal functions in laboratory tests within four weeks before the registration.

  * Leukocyte count ≥ 3,000/μL
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 7.5 × 10^4/μL
  * Serum creatine level ≤ 3.0 mg/dL
  * 8.5 mg/dL ≤ corrected serum level of calcium ≤ 11.5 mg/dL
  * Total bilirubin ≤ 1.8 mg/dL
  * Aspartate aminotransferase (AST) Levels ≤ 90 IU/L
  * Alanine aminotransferase (ALT) Levels ≤ 100 IU/L
  * Patients who agreed to participate in this clinical study in writing after receiving sufficient explanation

Exclusion criteria:

* Patients with poorly-controlled dental caries
* Patients with double cancer that requires treatment
* Patients who are using following steroid drugs (except for topical ointment)
* Patients with poorly-controlled hypertension or cardiovascular disease
* Patients with active infectious diseases or HIV or hepatitis virus infections
* Other patients whose participation in the present study is considered inappropriate by a Principal Investigator or Clinical Investigator

PRIOR CONCURRENT THERAPY:

* No prior androgen-blockade therapy
* No prior or other concurrent anticancer therapy
* No prior or concurrent immunologic adjuvant therapy
* No prior or concurrent steroid drugs (except ointment)
* No other prior or concurrent bisphosphonates (excluding zoledronic acid)
* No prior systemic chemotherapy

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | 6 years
  The interval from the date of randomization to the earliest date on which prostate-specific antigen (PSA) progression, clinical progression, first skeletal-related events (SRE), death, or cessation of protocol treatment for any reason occurred.

SECONDARY OUTCOMES:
Time to first skeletal-related events (SRE) | 6 years
  The interval from the date of randomization to the earliest date of the first SRE or death for any reason. But exlude tha another SRE existing case on the same region as of the randomization.
Overall survival | 6 years
  The interval from the date of randomization to death for any reason.
Extent of disease on bone scan (EOD) | Baseline, Month 12, 24 and 36
  Ransition of EOD bone scan grade at randomization, 12, 24, 36 months after the therapy.
Pain scale | Baseline, Month 12, 24 and 36
  Ransition of with/without narcotic drug usage at randomization, 12, 24, 36 months after the therapy and if the case of without usage, ransition of rest pain scale.
FACES pain-rating scale | Baseline, Month 12, 24 and 36
  Ransition of FACES pain-rating scale at randomization, 12, 24, 36 months after the therapy.
Adverse events | Month 6, 12, 18, 24 and 30
  Adverse events from date of starting protocol treatment until 28 days after date of finishing the treatment are evaluated according to Japanese version of the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) by Translational Research Informatics Center.
QOL (SF-36) | Month 6, 12, 18, 24, 30 and 36
  Rantision of QOL health survey scale durintg protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Ogawa, MD, Ph.D., Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906